CLINICAL TRIAL: NCT03884153
Title: Selective Depletion of C-reactive Protein (CRP) With Therapeutic Apheresis (CRP Apheresis) in Stroke
Brief Title: CASTRO-B - Study on CRP Apheresis in STROke Patients in Berlin
Acronym: CASTRO-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other); Department of Nephrology and Internal Intensive Care Medicine, Charite, Berlin (Unknown)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASTRO-B
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Stroke, Ischemic
Keywords: Ischemic Stroke; CRP apheresis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Comparisons will be drawn from historic controls from previous observational stroke studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRP apheresis (Experimental): CRP apheresis by means of selective apheresis using the "PentraSorb"-CRP adsorber
  Interventions: Device: CRP apheresis

INTERVENTIONS:
Device: CRP apheresis — selective CRP apheresis by use of the "PentraSorb"-CRP

SUMMARY:
This study explores the use of CRP level reduction in patients after suffering from acute ischemic stroke. Using selective CRP-apheresis, the investigators aim to reduce the secondary inflammatory tissue damage in the course of infarction maturation using infarction growth in MRI as the primary outcome as a surrogate.

DETAILED DESCRIPTION:
C-reactive protein (CRP) is an acute-phase protein binding to phosphocholine, thereby marking damaged tissue. This in turn activates the complement system and the cellular immune system engaging the unspecific immune system in an inflammatory tissue-degrading reaction. Such a pattern is observed in ischemic stroke, and elevated CRP levels can be measured in stroke survivors' sera. Several observational studies reproduced higher CRP levels with negative outcome in stroke. In another vascular model disease, myocardial infarction, selective CRP apheresis reduced infarct size in humans. The investigators therefore designed this pilot study to explore the effects of selective CRP reduction in ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years
* Informed consent signed by patient
* Patients with acute ischemic stroke in the Arteria cerebri media (MCA) territory within 36 hours of event
* Acute MRI with evidence of infarction
* NIHSS ≥ 4
* CRP > 5 mg/l

Exclusion Criteria:

* Withdrawal of consent
* Systolic blood pressure <100 mmHg before the apheresis
* Blood pressure relevant extra- and intracranial stenoses (NASCET 70)
* Apheresis contraindication
* Participation in other interventional studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Infarct growth | 5 ± 1 days after infarction
  Infarct growth measured via DWI-FLAIR volume change

SECONDARY OUTCOMES:
Infarct growth | 90 ± 14 days after infarction
  Infarct growth measured via diffusion-weighted imaging (DWI)-FLAIR volume change
Stroke Severity | 5 ± 1 days after infarction
  National Institute of Health Stroke Scale (NIHSS) score - ranging from 0-42 - higher values represent a worse outcome
Functional Outcome | 90 ± 14 days after infarction
  Modified ranking scale (mRS) score - ranging from 0-6 with higher scores signifying worse outcome no subscales
Dependency | 90 ± 14 days after infarction
  Barthel Index (BI) - ranging from 0-100 with higher scores signifying better outcome; no subscales
Cognitive Impairment | 90 ± 14 days after infarction
  Montreal Cognitive Assessment (MoCA) - ranging from 0-30 with higher scores signifying better outcome; no subscales
Quality of Life after Stroke via Stroke Impact Scale (SIS) | 90 ± 14 days after infarction
  Stroke Impact Scale - Stroke Impact Scale (SIS) - measures different aspects of the overall impact of stroke on the patients' health and quality of life with different subscales addressing different domains:
  * physical problems
  * memory and thinking
  * mood and emotions
  * communication
  * daily activities
  * mobility
  * motor impairment hand
  * participation
  * overall recovery higher values represent better outcome
Incidence of Complications | 90 ± 14 days after infarction
  Composite frequency of Complications within the time frame

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Zentrum für Schlaganfallforschung (CSB) / Klinik für Neurologie mit Experimenteller Neurologie der Charité, Berlin, Germany